CLINICAL TRIAL: NCT02674347
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Escalating Doses of Intravenous Zidebactam in Healthy Adult Human Subjects
Brief Title: MAD Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Intravenous Zidebactam in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: W-5107-102
Record Dates: First submitted 2016-01-25; First posted 2016-02-04 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — zidebactam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: 3 g or 6 g of Zidebactam (Experimental): Cohort 1 (Zidebactam): 3 g of Zidebactam (1 g every 8 hours [q8h]) (n=8) IV infusions administered over 60 minutes.
  Cohort 2 (Zidebactam or placebo): 6 g of Zidebactam (2 g q8h) (n=8) IV infusions administered over 60 minutes.
  Interventions: Drug: 3 g or 6 g Zidebactam
- Placebo (Placebo Comparator): Cohort 1: Placebo every 8 hours [q8h] (n=2) IV infusions administered over 60 minutes.
  Cohort 2: Placebo every q8h (n=2) IV infusions administered over 60 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3 g or 6 g Zidebactam — IV for over a duration of 60 minutes
  Other Names: WCK 5107
  Arms: Cohort 1: 3 g or 6 g of Zidebactam
Drug: Placebo — IV matching the Investigational drug
  Arms: Placebo

SUMMARY:
Study to evaluate the safety and tolerability of multiple escalating doses of intravenous (IV) Zidebactam in healthy adult human subjects.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled study where healthy adult subjects will be randomly assigned to receive either of the investigational products (Zidebactam or placebo) in 2 multiple ascending dose (MAD) cohorts.

Primary Objective: to evaluate the safety and tolerability of multiple escalating doses of intravenous (IV) zidebactam in healthy adult human subjects.

Secondary Objective: to evaluate the pharmacokinetics (PK) of multiple escalating doses of IV zidebactam in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have a body mass index of 18 to 30 kg/m2 (both inclusive) calculated as weight (kg)/height (m2).
2. Medical history without any major pathology/surgery in the last 6 months prior to screening.
3. All values of hematology, serum chemistry, coagulation, and urinalysis showing no clinically significant deviations from normal as judged by the Principal Investigator.
4. Resting supine blood pressure of 90 to 139 (systolic)/40 to 89 (diastolic) mmHg and a resting pulse rate of 40 to 100 beats per minute.
5. Calculated creatinine clearance ≥80 mL/min (Cockcroft-Gault method).
6. Computerized 12-lead ECG recording without signs of clinically significant pathology and showing no clinically significant deviation as judged by the Principal Investigator.

Exclusion Criteria:

1. History of clinically significant food or drug allergy, including known hypersensitivity to β lactam drugs or other related drugs.
2. History of Clostridium difficile induced diarrhea or infection within 1 year before screening
3. Consumed more than 28 units of alcohol per week at any time in the 6 months before investigational product administration
4. History/evidence of clinically relevant pathology related to the cardiovascular system, central nervous system, respiratory tract, gastrointestinal tract, endocrinology, immunology, hematology or any other systemic disorder/major surgeries, that in the opinion of the Principal Investigator would confound the subject's participation and follow-up in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated by reported AEs, clinical observations, vital signs measurements, and physical examination findings. | 14 days
Safety and tolerability will be evaluated by 12-lead safety ECG results and clinical laboratory test results | 14 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters -maximum plasma concentration will be evaluated. | 7 days
Pharmacokinetic parameters- area under the plasma concentration-time curve from zero (pre-dose) to 8 hours will be evaluated. | 7 days
Pharmacokinetic parameters- terminal half life etc will be evaluated | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No